CLINICAL TRIAL: NCT02961920
Title: The Influence of Prolonged Inspiratory Time on Respiratory Mechanics and Oxygenation in Obese Patients Undergoing Spine Surgery in the Prone Position
Brief Title: The Effect of Prolonged Inspiratory Time on Pulmonary Mechanics in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Jung Ju Choi, assistance professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PrIspSp
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Results first posted 2019-10-07 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IE ratio 1:1 (Experimental): Set an I(inspiration):E(expiration) ratio1:1 in the mechanical ventilator during spine surgery in the prone position in obese patients.
  Interventions: Device: IE ratio 1:1
- IE ratio 1:2 (Active Comparator): Set an I(inspiration):E(expiration) ratio1:2 in the mechanical ventilator during spine surgery in the prone position in obese patients.
  Interventions: Device: IE ratio 1:2

INTERVENTIONS:
Device: IE ratio 1:1 — Set an I:E ratio1:1 in the mechanical ventilator during spine surgery in the prone position in obese patients.
  Other Names: one and one
  Arms: IE ratio 1:1
Device: IE ratio 1:2 — Set an I:E ratio1:2 in the mechanical ventilator during spine surgery in the prone position in obese patients.
  Other Names: one and two
  Arms: IE ratio 1:2

SUMMARY:
The area of aesthesia-induced atelectasis is much larger in the obese compared with the non-obese, but there may also be more airway closure and impaired matching of ventilation and lung blood flow.

When an anesthetized patient is turned to the prone position, dynamic compliance (Cdyn) decreases and peak airway pressure increases unless the abdomen hangs freely to prevent the abdominal viscera from compromising the diaphragm movement. Although the Wilson frame is designed to allow the abdomen to hang, it partially compresses the anterior abdominal wall and therefore does not allow the abdomen to hang completely, especially in obese patients.

This in turn increases peak airway pressure and decreases Cdyn, oxygenation. This study aimed to investigate the effects of a prolonged I:E ratio (i.e., 1:1) compared with the conventional I:E ratio of 1:2 on respiratory mechanics and hemodynamics during spine surgery in the prone position in obese patients.

We hypothesized that, compared with an I:E ratio of 1:2, a ratio of 1:1 improve oxygenation without hemodynamic instability .

DETAILED DESCRIPTION:
After written informed consent was obtained from all patients, 50 adult patients were enrolled in the study.

The patients met the following inclusion criteria: (1) body mass index (BMI, weight in kilograms divided by the square of height in metres) > 25 kg/m2; (2) American Society of Anesthesiology (ASA) physical status classification grade I or II (BMI by itself was not used as the basis for the ASA classification); (3) aged 20 - 65 years; and (4) scheduled for elective spine surgery in prone position.

Exclusion Criteria:

* Patients who have severe pulmonary disease:

history of chronic obstructive pulmonary disease (COPD), asthma, or pneumothorax. Patients with haemodynamic instability, hypovolaemia, bronchopleural fistula, The enrolled patients were randomly allocated according to a predetermined allocation sequence to receive an I:E ratio of either 1:1 (group 1:1) or 1:2 (group 1:2).

The allocation sequence with no blocking was generated in an Internet website Standard monitoring techniques, including electrocardiography, pulse oximetry, and noninvasive arterial blood pressure measurement, are applied upon arrival at the operating room.

Anesthesia was induced with intravenous propofol 1.5 mg_kg-1 and rocuronium 0.8 mg_kg-1 was administered intravenously.

After tracheal intubation, volume-controlled ventilation was initiated with an I:E ratio of 1:2 or 1:1, no positive end-expiratory pressure, and a tidal volume of 10 mL per ideal body weight (kg). A respiratory rate was adjusted in order to end-tidal carbon dioxide (EtCO2) of 33 - 36 mmHg during surgery. Anesthesia was maintained with an end-tidal concentration of 2-2.5 vol% sevoflurane in 40% oxygen/air. The bispectral index score was monitored continuously in order to maintain an adequate anesthetic depth and was targeted at a range of 40-60 during surgery.

Radial artery cannulation was conducted for monitoring continuous arterial blood pressure and blood sampling.

Respiratory, hemodynamic, and arterial blood gas data were assessed and recorded at three time points: ten minutes after tracheal intubation in the supine position (T1), 30 min after prone positioning (T2), 90 min after prone positioning(T3). Respiratory data consisted of peak airway pressure, plateau airway pressure, mean airway pressure, static compliance, EtCO2, respiratory rate, and minute volume. Arterial pH, arterial oxygen tension (PaO2), arterial carbon dioxide tension (PaCO2), and lactate level were obtained from arterial blood gas analysis.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II adult patients scheduled for spine surgery under general anesthesia.
* patient age : greater than 20 years and less than 65years
* Body Mass Index(BMI) >25 kg/m2

Exclusion Criteria:

* Patients who have severe pulmonary disease:

history of chronic obstructive pulmonary disease (COPD), asthma, or pneumothorax. Patients with haemodynamic instability, hypovolaemia, bronchopleural fistula, history of cardiopulmonary disease, or previous lung surgery are excluded.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Cheon Lee, MD, Study Chair — Gachon University Gil Medical Center
Locations (1):
- Kyung Cheon Lee, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2016 and October 2018, 50 patients who underwent lumbar spine surgery in our institution were assessed. Two patients dropped out. Thus, 48 patients achieved study protocol.
Period: Overall Study
Arm/Group | IE Ratio 1:2 | IE Ratio 1:1
Started | 25 | 25
Completed | 24 | 24
Not Completed | 1 | 1
Not completed — did not achive stydy protocol schedule | 1 | 1

BASELINE CHARACTERISTICS:
Population: did not achieve stydy portocol schedule 2
Groups:
- Total: Total of all reporting groups
Arm/Group | IE Ratio 1:1 | IE Ratio 1:2 | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 48
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (10) | 54.6 (13) | 53.42 (9.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 18 | 13 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 24 | 24 | 48
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 24 | 24 | 48
body mass index [Mean (Standard Deviation); unit: kg/m^2] | 27.4 (7.9) | 28.7 (2.7) | 28.13 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: PaO2(Partial Pressure of Oxygen in Arterial Blood)
Description: ten minutes after tracheal intubation to 90 min after prone position
Time Frame: ten minutes after tracheal intubation to 90 min after prone position
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | IE Ratio 1:2 | IE Ratio 1:1
Number analyzed (Participants) | 24 | 24
mmHg
  paO2 30min | 178.71 (36.43) | 198.04 (17.667)
  PaO2 90min | 185.25 (26.54) | 202.54 (17.627)

ADVERSE EVENTS:
Time Frame: 7days
Description: desaturation We checked daily O2 saturation and if the saturation below 90% then we define as desaturation.
Arm/Group | IE Ratio 1:2 | IE Ratio 1:1
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT02961920/Prot_SAP_000.pdf